CLINICAL TRIAL: NCT03655028
Title: Increasing Physical Activity in COPD Through Rhythmically Enhanced Music
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2803-R
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: COPD Patients and Patients Recovering From COVID19
Keywords: COPD; Exercise; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial in which COPD patients in the intervention group and COVID19 patient in the intervention group will undergo a home-based, exercise program augmented with RAS-enhanced music while COPD patients in the control group and COVID19 patients in the control group will undergo a home-based, exercise program without music. Outcomes of the home-based exercise program with music will be compared to the outcomes of home-based exercise alone. Outcomes are listed below.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both investigator and outcome assessor will be blinded to patient allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RAS-music group (Experimental): Home-based, exercise program augmented with rhythmically auditory stimulation enhanced music
  Interventions: Behavioral: rhythmically auditory stimulation enhanced music
- Control group (Active Comparator): Home-based, exercise program without rhythmically auditory stimulation enhanced music
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: rhythmically auditory stimulation enhanced music — Patients in the intervention group will listen to music enhanced by rhythmic auditory stimulation while engaging in a 12-week home-based exercise program
  Arms: RAS-music group
Behavioral: control — Patients in the control group will not listen to music while engaging in a 12-week home-based exercise program
  Arms: Control group

SUMMARY:
The VA cares for nearly one million Veterans with COPD at a cost of more than $5.5 billion annually. COPD profoundly impairs quality of life as it limits ability to work, to maintain physical exertion and to engage in social activities. Hospital-based rehab can decrease the need for inpatient and outpatient medical care and can improve exercise capacity, quality of life and, possibly, decrease mortality. Unfortunately, access to hospital-based VA rehab is insufficient and, over time, the few Veterans who attend experience progressive loss of functional gains. The investigators reason that the proposed home-based exercise program augmented by patient-tailored, RAS-enhanced music will overcome the many limitations of hospital-based rehab. Through this innovative program, the investigators expect to enhance the benefits of rehab and better maintain them over time. The easy applicability of this innovative, accessible and economical program has the potential to modify the spiraling pattern of increasing disability and reduce health-care cost and mortality in Veterans with COPD.

In 2021, the investigators obtained an 'Administrative Project Modification' to the parent COPD study in which they will include patients recovering from prolonged COVID19 hospitalization. Specifically, the investigators will use the novel RAS-enhanced music exercise program developed for the parent grant in patients recovering from COVID19. The main goal of the modified proposal for COVID19 patients will be to compare the efficacy of a 12-week, home-based exercise program augmented by RAS-therapeutic music and strength training to 12-weeks usual care and strength training in patients recovering from COVID 19.

DETAILED DESCRIPTION:
Rationale: In COPD, hospital-based pulmonary rehabilitation can improve symptoms, functional status, and quality of life and decrease unscheduled physician visits, emergency room visits, hospitalizations, and possibly, mortality. Despite the well documented efficacy, hospital-based rehab remains inadequate due to insufficient access, acceptance and sustainability. This has triggered a growing interest in home-based rehab programs. Patients enrolled in home-based programs, however, may exercise at low intensities to avoid dyspnea/fatigue, limiting the potential benefits of exercise training. Accordingly, it is essential to develop innovative home-based programs that decrease exercise-induced dyspnea and fatigue while ensuring sufficient exercise intensity to produce sustainable physiologic benefit. Recent data suggest that rhythmically auditory stimulation (RAS) using music may constitute such an innovative strategy. Music can diminish exercise-induced dyspnea/fatigue allowing patients to tolerate more challenging physical activity and obtain a greater benefit from rehab. Music also can induce entrainment of motor responses such as walking. The investigators thus plan to capitalize on both the sensorimotor coupling of gait with RAS-enhanced music and the mitigating effect of music over exercise-induced dyspnea/fatigue. Specifically, the investigators propose to compare the efficacy of a 12-week, home-based exercise program augmented by patient-tailored, RAS-enhanced music to a 12-week traditional home-based exercise program in patients with COPD. Hypothesis: (H1) Compared to patients randomized to a home-based, exercise program without music (control group), patients randomized to a home-based, exercise program augmented with RAS-enhanced music (intervention group) will demonstrate (H1a, primary hypothesis) greater increase in 6-minute walk distance, (H1b) greater increase in walking time on a constant-load treadmill test protocol, (H1c) reduced dyspnea during a constant-load treadmill test protocol, and (H1d) greater increases in health-related quality of life. In addition (H2), they will accumulate greater volume of physical activity (actigraphy) and (H3) will better sustain these benefits over time. Lastly (Explorative Objective), the investigators will assess the mechanistic impact physiological and psychological phenotype and clinical factors on responsiveness to rehabilitation (duration constant-load treadmill test) achieved with and without concurrent use of RAS-music. Methods: The proposed study is a randomized, controlled clinical trial in which 170 patients will be randomized into a home-based, exercise program without music or a home-based exercise program augmented with RAS-enhanced music. Patients will receive 12-weeks of home-based training per group assignment (at least three times weekly) followed by 12-weeks of follow-up to assess the sustainability of the investigators' novel intervention. Testing will be carried out at baseline and at 6, 12 and 24 weeks. Testing will include pulmonary function test, 6-minute walk tests, constant-load treadmill test, physical activity quantification, measurements of dyspnea, quality of life, and objective quantification of quadriceps dimensions (ultrasonography) and strength/fatigue (magnetic stimulation of the femoral nerve). Analysis: In the principal analysis of the primary outcome measure (6-minute walk distance) the investigators will use a mixed-model analysis that includes, treatment, time and treatment-by-time interaction terms. This model will automatically account for missing data-where missing at random is assumed. The investigators will conduct a sensitivity analysis based on the results of the mixed model analysis to determine which other assumptions regarding missing data might produce different results. One component of the sensitivity analysis will include adjustment for baseline demographic and health covariates. A linear regression model and a mixed model ANOVA will be used to assess the impact of clinical confounders (Explorative Objective). Scientific contribution: These data will provide a solid foundation to determine the physiologic impact of the rehab strategy. This innovative, practical and economical pulmonary rehabilitation strategy has the potential to create a paradigm shift in the care of the many Veterans with COPD who have no access to pulmonary rehabilitation. The above-described protocol will be also tested in patients recovering form COVID19. The investigators reason that the proposed innovative, practical, safe and economical program has the potential to create a paradigm shift in the care of the many veterans who were hospitalized with COVID19 and who have no access to physical rehabilitation.

Please note: Due to the COVID-19 pandemic, constant load treadmill testing could not be completed as was originally proposed. There was concern that COVID-19 could be transmitted due to increased exposure to increased saliva associated with testing. Therefore, the objectives using constant load testing will not be reported. The exploratory objective was based on the constant workload treadmill test so that is not reported. Additionally, again due to the COVID-19 pandemic, 6-week testing was not completed after the pandemic due to the increased risk of transmission (n.b., 6-week data were not included in the outcomes and was to be used for analysis of the primary objective; as such, the analysis of the primary objective was changed to ANCOVA from what was in the protocol). The protocol attached here is the last approved IRB protocol and includes both patients with COPD and COVID. Only data on patients with COPD are reported here. The two groups of patients were two different populations and it does not make theoretical sense to combine the data at this point. Text concerning COVID are in gray.

ELIGIBILITY:
Inclusion Criteria:

COPD patients:

* =< 40 yr. of age
* FEV1 =< 70%
* FEV1/FVC <70%
* Mean SpO2 88% at peak exercise (with or without oxygen supplementation)

COVID19 patients

* >=18 yrs. of age
* Previous hospital and/or emergency room visit for laboratory-confirmed COVID-19 diagnosis.
* Able to walk independently
* Mean SpO2 88% at peak exercise (with or without oxygen supplementation)
* Ability to hear music

Exclusion Criteria:

COPD patients:

* Respiratory infection/COPD exacerbation within the previous four weeks
* Exercise-limiting heart disease

  * Congestive heart failure - i.e., New York Heart Association Class III or IV
  * Positive stress test or other indicators of heart disease or complaints of angina during the stress test
* Exercise-limiting peripheral arterial disease

  * Stops walking due to intermittent claudication
* Stops exercise for arthritic pain in knee or hips
* Inability to walk on the treadmill
* Any unforeseen illness or disability that would preclude exercise testing or training
* Participation in a formal exercise program within the previous 12-weeks

COVID patients:

* Able to walk more than 550 meters during a standard 6-minute walk test
* Exercise limiting heart disease

  * Complaints of angina during the 6- minute walk distance tests or other indicators of exercise-limiting heart disease
* Congestive heart failure (New York Heart Association Class III or IV)
* Exercise-limiting peripheral arterial disease (stops exercise due to intermittent claudication)
* Stops exercise due to arthritic pain in the knee or hips (self-report)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Laghi, MD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 93 participants met the criteria and were randomized into the study.
Period: Baseline
Arm/Group | RAS-music Group | Control Group
Started | 46 | 47
Completed | 46 | 47
Not Completed | 0 | 0
Period: 12-weeks Follow up
Arm/Group | RAS-music Group | Control Group
Started | 46 | 47
Completed | 36 | 40
Not Completed | 10 | 7
Not completed — Death | 1 | 0
Not completed — Physician Decision | 3 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 4 | 4
Period: 24-weeks
Arm/Group | RAS-music Group | Control Group
Started | 36 | 40
Completed | 35 | 38
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Music plus 12-week walking program
- Control: 12-week walking program only
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 14
  >=65 years | 36 | 43 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (6) | 73 (6) | 71 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 7
  Male | 39 | 47 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 45 | 45 | 90
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 9 | 25
  White | 30 | 38 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 47 | 93
FEV1 [Mean (Standard Deviation); unit: Liters] — Forced expiratory volume in 1 second
  Liters | 1.49 (.51) | 1.39 (.46) | 1.44 (.49)
FEV1 percent predicted [Mean (Standard Deviation); unit: percent predicted] | 48 (13) | 45 (15) | 47 (14)
FEV1/FVC [Mean (Standard Deviation); unit: percent] | 51 (11) | 47 (13) | 49 (12)
Six minute walk distance [Mean (Standard Deviation); unit: meters] | 433 (81) | 403 (98) | 418 (91)
Dyspnea [Mean (Standard Deviation); unit: units on scale] — Scale range from 0-10; with 0 = none and 10= max dyspnea
  units on scale | 3.4 (1.9) | 3.5 (1.6) | 3.5 (1.7)
Daily step count [Mean (Standard Deviation); unit: steps per day] | 3308 (1346) | 2750 (1648) | 3008 (1532)

OUTCOME MEASURES:

1. Primary Outcome: Six-minute Walk Distance
Description: Patients will be instructed to walk as fast as they can without running for six minutes. The test will be conducted according to ATS standards. Distance will be recorded in meters walked. Outcomes will be compared between the intervention groups.
Time Frame: 12 weeks
Population: Participants assigned to each group who completed 12-week testing
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 40
meters | 452 (79) | 429 (105)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.85, ANCOVA — The co-variate used in the analysis was the 6 minute walk distance at baseline

2. Secondary Outcome: Volume of Daily Physical Activity
Description: Volume of daily physical activity over a seven day period will be recorded using a triaxial accelerometer worn on the hip (actigraph). Volume of physical activity will be compared between the intervention group and the control group.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 40
steps per day | 3930 (2551) | 3738 (2566)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = .307, ANCOVA — The co-variant used to adjust the ANCOVA was the baseline step count/day

3. Secondary Outcome: Six-minute Walk Distance
Description: To determine whether, 24-weeks after randomization, gains in 6-minute walk distance and perceived functional improvements will be sustained to a greater extent in the rhythmic auditory stimulation enhanced music group than in the control group the six-minutes walk test will be repeated 24-weeks after randomization. During the six-minute walk test patients will be instructed to walk as fast as they can without running for six minutes. The test will be conducted according to ATS standards. Distance will be recorded in meters walked. Outcomes will be compared between the two groups.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Intervention | Control
Number analyzed (Participants) | 35 | 38
meters | 444 (82) | 439 (107)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.106, ANCOVA — this comparison is made between distance walked during 6MW at 12 weeks and distance walked during 6MW at 24 weeks

4. Secondary Outcome: Quality of Life Physical Function
Description: measured by the Short Form-36 Physical component score. Scores range from 0-100 (higher scores are better).
Time Frame: 12 weeks
Population: numbers of subjects are inconsistent because subjects did not complete the questionnaires
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: 12-week walking program onl
Arm/Group | Intervention | Control
Number analyzed (Participants) | 33 | 39
score on a scale | 40.4 (6.0) | 38.7 (7.3)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.26, ANCOVA — Baseline PCS score was used at the co-variate

5. Secondary Outcome: Quality of Life Mental Health
Description: Quality of Life measured by Short Form-36 Mental Component Scale (range=0-100; higher score is better)
Time Frame: 12-weeks
Population: some subjects did not complete the questionnaires
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: 12-week walking program
Arm/Group | Intervention | Control
Number analyzed (Participants) | 33 | 39
score on a scale | 42.8 (6.1) | 42.3 (6.6)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.85, ANCOVA — Covariate was baseline MCS score

6. Other Pre Specified Outcome: Adherence to Training Sessions Protocol
Description: number of walking exercise sessions completed
Time Frame: 12 weeks
Population: total number of sessions completed
Measure: Mean (Standard Deviation); unit: number of training sessions completed
Arm/Group | Intervention | Control
Number analyzed (Participants) | 36 | 40
number of training sessions completed | 25.6 (10.7) | 19.7 (12.8)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.025, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events are reported from randomization to study completion (typically 6-8 months)
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 1/46 | 1/47
Serious Adverse Events (participants affected / at risk) | 3/46 | 4/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=46) | Control (N=47)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) — Hospitalized for COPD exacerbation/pneumonia
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — pulmonary embolism hospitalization

LIMITATIONS AND CAVEATS:
The study was interrupted by the COVID-19 pandemic. Initially we were going to analyze data generated from metabolic stress testing. Due to the large amounts of saliva produced from these measures, we dropped metabolic stress testing from the protocol and substituted data generated from the 6MW test instead. Less subjects were enrolled than planned also due to the pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT03655028/Prot_SAP_000.pdf